CLINICAL TRIAL: NCT05009771
Title: Postoperative Pain Management of Caesarean Section: a Prospective, Observational Cohort Study
Brief Title: Postoperative Pain Management of Caesarean Section
Status: Recruiting | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chi-Hsu Wang, Principal Investigator, Mackay Memorial Hospital
Other Study IDs: 21MMHIS203e
Record Dates: First submitted 2021-08-03; First posted 2021-08-18 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; Caesarean Section; Analgesia
Keywords: Postoperative Pain; Caesarean section; Postpartum rehabilitation; Dinalbuphine sebacate; PCA; NALDEBAIN
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IV-PCA + NALDEBAIN group: Patients treated with the combination of IV-PCA and intramuscular injection of dinalbuphine sebacate will be allocated to IV-PCA + NALDEBAIN group.
  Interventions: Drug: Intravenous patient-control analgesia; Drug: Dinalbuphine sebacate
- IV-PCA group: Patients receiving intravenous patient-controlled analgesia (IV-PCA) will be allocated to IV-PCA group.
  Interventions: Drug: Intravenous patient-control analgesia

INTERVENTIONS:
Drug: Intravenous patient-control analgesia — At the two trial sites, IV-PCA is commonly used with morphine. The device is installed after delivery and removed within 3 days.
  Other Names: IV-PCA
Drug: Dinalbuphine sebacate — Dinalbuphine sebacate is a prodrug of nalbuphine. With oil-based formulation, the active ingredient releases slowly and the effect lasts longer than nalbuphine. After delivery, a single 150 mg dose of dinalbuphine sebacate is administered intramuscularly.
  Other Names: NALDEBAIN
  Groups: IV-PCA + NALDEBAIN group

SUMMARY:
Caesarean section is one of the most frequent surgeries causing severe postoperative pain. Poor management of acute pain can contribute to postoperative complications, late recovery and the development of chronic pain. Moreover, it had been demonstrated that the intensity of postpartum pain is associated with depression. It is imperative to find out appropriate methods of postpartum pain alleviation. Currently, a lot of analgesic drugs and methods have been developed and used in clinical practice, such as patient-controlled analgesia, extended-release analgesics and multimodal analgesia. This prospective cohort study is aimed to investigate the outcome of each postoperative analgesic method used in caesarean section.

DETAILED DESCRIPTION:
This is a prospective, observational, cohort study. Patients undergoing elective caesarean section will be invited to the study. The written informed consent will be obtained prior to participation. After getting the written informed consent, data will be collected from medical records, questionnaires, patient diaries, visit records and telephone visit records. Through telephone visits, postpartum depression scale and postpartum chronic pain will be evaluated six weeks and three months after delivery. Demographic data, consumption of analgesics, analgesic methods, intensity of postoperative pain, complications, recovery time, score of depression scale will all be summarized. Numerical variables will be present with mean and standard deviation and categorical variables will be present with number and percentage.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20 to 40.
2. Planing to undergo caesarean section with spinal anesthesia.
3. Scheduled to undergo cesarean section between 37 and 40 weeks of gestation.
4. American Society of Anesthesiology Physical Class 1-2.
5. Planing to alleviate postoperative pain with intravenous patient-controlled analgesia or administration of NALDEBAIN.

Exclusion Criteria:

1. Not willing to provide informed consent.
2. Unable to receive opioids or NSAIDs due to contraindication.
3. Long-term use of opioids or drug abuse.
4. Suffering from chronic pain disease.
5. Having medical history of mental illnesses.
6. Diagnosed with Pre-eclampsia or eclampsia.
7. Diagnosed with gestational diabetes.
8. Unsuitable for participation judged by investigator.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study population is pregnant woman.
Study Population: Pregnant woman scheduled to have caesarean section within 30 days.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Postpartum pain intensity | Within 5 days after delivery
  Pain intensity is assessed by numerical rating scale (NRS) at least twice daily during hospital stay after delivery. NRS is a 11-point scale which labeled from zero (no pain) to ten (worst pain). The area under the curve of NRS are calculated.

SECONDARY OUTCOMES:
Consumption of analgesics | Within 5 days after delivery
  The mean total consumption of analgesics during the hospital stay after delivery.
Incidence of complications | Up to 5 days after delivery
  the incidence of postoperative complication occurring during hospital stay after delivery, especially the ones related to analgesics.
Ambulation | Up to 5 days after delivery
  The mean length of time between delivery and the first ambulation.
Breastfeeding | Up to 5 days after delivery
  The percentage of participants able to breastfeed during hospital stay and the mean length of time between delivery and the first breastfeeding.
Gastrointestinal function recovery | Up to 5 days after delivery
  The mean length of time between delivery and first soft diet.
Postnatal Depression assessment | At baseline, 6 weeks and 3 months after delivery
  Edinburgh Postnatal Depression questionnaire is used to assess patients' postpartum depression. Participants are asked to fill in the questionnaire at baseline (within 30 days prior to delivery), 6 weeks and 3 months after delivery.
Satisfaction assessed by a four-point scale | 6 weeks after delivery
  Participants are asked to assess the satisfaction toward rate of recovery progress and pain management through 6 questions six weeks after delivery. Each question contain 4 choices: very satisfied, satisfied, dissatisfied and very dissatisfied.
Chronic pain intensity | 6 weeks and 3 months after delivery
  Chronic pain intensity is assessed by NRS 6 weeks and 3 months after delivery. NRS is a 11-point scale which labeled from zero (no pain) to ten (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hsu Wang, M.D., Principal Investigator — MacKay Memorial Hospital Tamsui Branch
Locations (2):
- Taiwan (2):
  - MacKay Memorial Hospital Tamsui Branch, New Taipei City, Taiwan
  - MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No